CLINICAL TRIAL: NCT07340853
Title: A Phase 1b Clinical Trial of CRISPR Delivered Anti-BCMA Chimeric Antigen Receptor T Cells for Treatment of Relapsed or Refractory Multiple Myeloma
Brief Title: CRISPR Delivered Anti-BCMA Car-T Therapy for Relapsed or Refractory Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Martin, MD (Other)
Responsible Party: Sponsor-Investigator, Thomas Martin, MD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25707; NCI-2025-08425 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma; Recurrent Multiple Myeloma; Refractory Multiple Myeloma
Keywords: CAR T; CRISPR
MeSH Terms: conditions — Multiple Myeloma | interventions — Leukapheresis; Cyclophosphamide; Immunotherapy, Adoptive; Quality of Life; Surveys and Questionnaires; Biopsy; Specimen Handling; fludarabine; Phantoms, Imaging; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation Starting Dose: 10 × 10^6 CAR + T cells/ infusion (Experimental): Participants undergo leukapheresis and then receive lymphodepleting chemotherapy with fludarabine IV over 30 minutes and cyclophosphamide IV over 60 minutes on days -5, -4, and -3. Participants also receive 10 × 10^6 BCMA CAR-T cells/ infusion over 5-30 minutes on day 1 in the absence of disease progression or unacceptable toxicity. Additionally, participants undergo PET/CT or MRI at screening and urine and blood sample collection, bone marrow biopsy or aspiration throughout the study.
  Interventions: Procedure: Leukapheresis; Drug: Cyclophosphamide; Biological: Chimeric Antigen Receptor T cells (CAR-T) Targeting BCMA; Behavioral: Quality of Life (QoL) Questionnaires; Procedure: Bone Marrow Biopsy; Biological: Biospecimen Collection; Drug: Fludarabine; Procedure: Radiographic imaging
- Dose Escalation: Planned Dose: 30 × 10^6 CAR + T cells/ infusion (Experimental): Dependent on the safety profile of the starting dose, participants undergo leukapheresis and then receive lymphodepleting chemotherapy with fludarabine IV over 30 minutes and cyclophosphamide IV over 60 minutes on days -5, -4, and -3. Participants also receive 30 × 10^6 BCMA CAR-T cells/ infusion over 5-30 minutes on day 1 in the absence of disease progression or unacceptable toxicity. Additionally, participants undergo PET/CT or MRI at screening and urine and blood sample collection, bone marrow biopsy or aspiration throughout the study.
  Interventions: Procedure: Leukapheresis; Drug: Cyclophosphamide; Biological: Chimeric Antigen Receptor T cells (CAR-T) Targeting BCMA; Behavioral: Quality of Life (QoL) Questionnaires; Procedure: Bone Marrow Biopsy; Biological: Biospecimen Collection; Drug: Fludarabine; Procedure: Radiographic imaging
- Expansion: MTD of Anti-BCMA CAR-T (Experimental): Participants undergo leukapheresis and then receive lymphodepleting chemotherapy with fludarabine IV over 30 minutes and cyclophosphamide IV over 60 minutes on days -5, -4, and -3. Participants also receive the MTD of BCMA CAR-T cells/ infusion established in the dose escalation phase over 5-30 minutes on day 1 in the absence of disease progression or unacceptable toxicity. Additionally, participants undergo PET/CT or MRI at screening and urine and blood sample collection, bone marrow biopsy or aspiration throughout the study.
  Interventions: Procedure: Leukapheresis; Drug: Cyclophosphamide; Biological: Chimeric Antigen Receptor T cells (CAR-T) Targeting BCMA; Behavioral: Quality of Life (QoL) Questionnaires; Procedure: Bone Marrow Biopsy; Biological: Biospecimen Collection; Drug: Fludarabine; Procedure: Radiographic imaging

INTERVENTIONS:
Procedure: Leukapheresis — Undergo Leukapheresis
Drug: Cyclophosphamide — Given Intravenously (IV)
  Other Names: Cycloblastin; Fosfaseron; Genoxal; Cytoxan
Biological: Chimeric Antigen Receptor T cells (CAR-T) Targeting BCMA — Given Intravenously (IV)
  Other Names: CAR-T Infusion
Behavioral: Quality of Life (QoL) Questionnaires — Ancillary studies
Procedure: Bone Marrow Biopsy — Undergo biopsy
  Other Names: Biopsy
Biological: Biospecimen Collection — Undergo Blood, serum and urine collection
  Other Names: Sample collection
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Radiographic imaging — Undergo radiographic imaging
  Other Names: Positron Emission Tomography (PET)/Computerized tomography (CT); PET/CT; Magnetic Resonance Imaging (MRI); MRI

SUMMARY:
This phase Ib trial tests the safety, side effects and best dose of clustered regularly interspaced short palindromic repeats (CRISPR) delivered anti-B-cell maturation antigen (BCMA) chimeric antigen receptor (CAR)-T cells (1XX BCMA CAR-T cells) in treating patients with multiple myeloma that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). Anti-BCMA CAR-T cell therapy is a type of treatment in which a person's T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein, such as BCMA, on the patient's cancer cells is added to the T cells in the laboratory by a tool called clustered regularly interspaced short palindromic repeats (CRISPR)-Cas9. The special receptor is called a CAR. Large numbers of the CAR-T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. Giving chemotherapy before CAR-T cells may decrease the number of lymphocytes (a type of white blood cells) in the blood and may help the 1XX BCMA CAR-T cells fight the cancer cells. Treatment with 1XX BCMA CAR-T cells may be safe, tolerable, and/or effective in treating patients with relapsed or refractory multiple myeloma (RRMM).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Dose Escalation:

I. To evaluate the safety and toxicity of administering Chimeric Antigen Receptor T Cells (CAR-T) cells targeting BCMA to participants with Relapsed or Refractory Multiple Myeloma (RRMM).

II. To determine the maximum tolerated dose (MTD) for anti-BCMA CAR-T cells.

Dose Expansion:

III. Determine whether administering conforming CAR T-cell product targeting BCMA to participants with RRMM increases the overall response rate (ORR) compared with historical data for non-CAR agents per International Myeloma Working Group (IMWG) response criteria.

IV. Determine whether administering conforming CAR T-cell product targeting BCMA to participants with RRMM lowers the Grade 2 or greater neurologic events to <10% in RRMM.

SECONDARY OBJECTIVES:

Dose Expansion:

I. To describe the efficacy of conforming CAR-T cell product targeting BCMA in participants with RRMM.

II. To evaluate the feasibility of manufacturing anti-BCMA CAR T-cells locally and ability to produce adequate quantities of vector positive T-cells.

III. To evaluate the safety and toxicity of conforming CAR-T cell product targeting BCMA to participants with RRMM.

EXPLORATORY OBJECTIVES:

I. To determine the degree and impact of CAR-T persistence following anti-BCMA CAR-T cell infusion, on clinical outcomes and safety.

II. Describe changes in health-related quality of life (HRQoL) using the European Organization for Research and Treatment of Cancer - Quality of Life C30 questionnaire (EORTC-QLQ-C30).

III. To describe the efficacy of CAR-T cells targeting BCMA in participants with relapsed or refractory BCMA+ RRMM who were treated with product that did not meet one or more pre-specified release criteria (non-conforming product cohort).

OUTLINE:

Participants in both cohorts will undergo leukapheresis, receive lymphodepleting chemotherapy and then receive a single infusion of BCMA CAR-T therapy. After completion of study treatment, participants are followed up at 30, 60 and 90 days, 6 and 12 months, and then yearly for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign informed consent form.
2. Age ≥18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
4. Diagnosis of multiple myeloma (per IMWG criteria) with relapsed or refractory disease and has received at least 3 prior lines of therapy including proteasome inhibitor immunomodulatory therapy, and anti-Cluster of differentiation 38 (CD38) antibody therapy.
5. Participants may have received BCMA targeted therapy and must be at least 6 months from last BCMA therapy.
6. Participants must have documented evidence of progressive disease within 12 months of the last line of therapy or be refractory/nonresponsive to their most recent line.
7. Participants must have measurable disease, defined as at least one of the criteria below:

   * Serum M-protein greater or equal to 0.5 grams per deciliter (g/dL).
   * Urine M-protein greater or equal to 200 milligrams, over a 24-hour period (mg/24 h).
   * Serum free light chain (FLC) assay: involved FLC level of ≥ 100 milligrams per liter (mg/L).
8. Adequate organ function, defined as:

   * Adequate bone marrow function for apheresis and lymphodepleting chemotherapy.
   * Hgb >8 gm/dl (transfusions allowed).
   * Platelets >50,000/microliter (uL) (in the absence of platelet transfusion within 7 days of apheresis, but transfusion permitted prior to lymphodepleting chemotherapy).
   * Absolute neutrophil count (ANC) > 1000/uL in the absence of growth factor support (filgrastim within 7 days or pegfilgrastim within 14 days of apheresis, but growth factor permitted prior to lymphodepleting chemotherapy). For those patients who have evidence of duffy null, ANC >750/uL is allowed.
   * Absolute lymphocyte count (ALC) >300/uL.
   * Alanine aminotransferase/aspartate aminotransferase (ALT/AST) < 3 x institutional upper limit of normal (ULN) and Total bilirubin < 1.5 milligrams per deciliter (mg/dl) x institutional ULN, except with Gilbert's syndrome.
   * Serum creatinine clearance (CrCl) ≥ 30 milliliter per minute (mL/min) using Cockcroft-Gault formula or as measured with a 24 hour urine collection.
   * Adequate cardiac function, defined as left ventricular ejection fraction (LVEF) > 40% as assessed by echocardiogram or multiple uptake gated acquisition (MUGA) and adequate pulmonary function (measured by room air pulse oximetry ≥ 92%).
9. Women of childbearing potential must have a negative serum or urine pregnancy test AND agree to use highly effective methods of contraception for 1 year after the last dose of anti-BCMA CAR-T cells.
10. Males who have partners of childbearing potential must agree to use an effective barrier contraceptive method for 6 months after CAR-T therapy.

Exclusion Criteria:

1. Autologous transplant within 12 weeks of planned CAR-T cell infusion.
2. Prior antitumor therapy as follows, prior to apheresis:

   * Investigational therapy within 14 days, or at least 5 half-lives.
   * Monoclonal antibody therapy within 21 days.
   * Cytotoxic therapy within 14 days.
   * Proteasome inhibitor therapy within 14 days.
   * Immunomodulatory therapy within 14 days.
   * Radiotherapy within 14 days - with the exception that if radiotherapy (XRT) covers <5% of marrow reserve - no rest window needed.
3. Toxicity from previous anticancer therapy must resolve to baseline levels or to Grade 1 or less except for alopecia, peripheral neuropathy and baseline hematologic toxicity that otherwise meets inclusion.
4. Active CNS multiple myeloma, plasma cell leukemia, primary AL amyloidosis or POEMS syndrome.
5. Active other malignancy, other than non-melanoma skin cancer, carcinoma in situ (e.g., cervix, bladder, or breast). Any fully treated malignancies or indolent, clinically insignificant malignancies can be discussed among the study team to determine eligibility.
6. HIV seropositivity.
7. Serologic status reflects active hepatitis B or C infection. Participants that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive participants will be excluded).
8. Participants with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, pulmonary abnormalities, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Pregnant or breastfeeding women are excluded from this study because CAR-T cell therapy may be associated with the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with CAR-T cells, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study.

   NOTE: Women of childbearing potential must have a negative serum or urine pregnancy test.
10. Participants with currently symptomatic central nervous system (CNS) pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia, and Parkinson's disease OR seizure or stroke within 6 months.
11. History of autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus) with requirement of immunosuppressive medication within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2028-05-25 (Estimated); Study Completion 2043-05-25 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with treatment-emergent adverse events | Up to 12 months following CAR-T infusion
  Proportion of participants with treatment-emergent adverse events of CAR-T in RRMM as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 5.0), revised Cytokine Release Syndrome (CRS) grading criteria (for CRS grading), and the American Society for Transplantation and Cell Transplantation (ASTCT) Immune effector cell-associated neurotoxicity syndrome (ICANS) Consensus Grading for Adults (for neurotoxicity grading).
Proportion of participants who experience dose-limiting toxicity (DLT) (Dose Escalation) | Up to 30 days
  The DLT evaluable analysis set includes all participants in the dose-finding part of the study who have received the target doses of anti-BCMA CAR-T cell product, and who have either experienced a DLT or were followed for the full DLT evaluation period. The trial observation period for dose limiting toxicities will conclude at day 30 (approximately 4 weeks after CAR-T cell infusion)
Maximum Tolerated Dose (MTD) (Dose Escalation) | Up to 28 days
  The DLT evaluable analysis set includes all participants in the dose-finding part of the study who have received the target doses of anti-BCMA CAR-T cell product, and who have either experienced a DLT or were followed for the full DLT evaluation period (within 28 days following infusion of CAR-T cells targeting BCMA). The MTD is defined as the dose level immediately below that in which ≥ 2/6 participants experience a DLT.
Best Overall Response Rate (BORR) (Dose expansion + MTD dose escalation cohort) | Up to 12 months following CAR-T infusion
  ORR is defined as the proportion of participants with stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), as per International Myeloma Working Group (IMWG) criteria, as best overall response over the total population. ORR will be reported as proportion with 90% binomial confidence interval for the expansion cohort including the patients on MTD in the dose escalation cohort(s).
Proportion of participants with of severe neurologic events (Dose Expansion) | From initiation of study treatment to 12 months following CAR-T infusion, approximately 13 months total
  Incidence of severe neurologic events defined as grade 2 or higher will be reported as a proportion of the total participants by group.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) - Long term | Up to 15 years
  The ORR from initiation of study treatment until disease progression or death from any cause will be reported as the proportion of participants with stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), as per International Myeloma Working Group (IMWG) criteria. ORR will be reported as proportion with 90% binomial confidence interval for each cohort
Median Duration of Response (DoR) - Beginning of response | Up to 15 years
  The median duration of response measured for responders, from the documented beginning of response ( sCR, CR, PR or VGPR) (as per IMWG criteria) until progression or death from any cause along with 95% confidence intervals.
Median Progression-free Survival from Study Entry (PFS-SE) | up to 15 years
  Progression-free Survival (PFS) is defined as the time from entry onto study until multiple myeloma progression or death from any cause. Where there is missing information, censoring of the data may be defined as the last date at which progression status was adequately assessed or the first date of unscheduled new anti-MM treatment and will be analyzed by Kaplan-Meier method for the expansion cohort including the participants on MTD in the dose escalation cohort.
Median DoR - First documented response | up to 15 years
  The median duration of response measured for responders is defined as the time from first response until multiple myeloma (MM) progression or death from any cause.
Median Overall Survival (OS) | up to 15 years
  The median overall survival is defined as the amount of time from study treatment until death and will be analyzed by Kaplan-Meier method for the expansion cohort including the participants on MTD in the dose escalation cohort.
Rates of MRD (-) and sustained MRD (-) | Up to 15 years
  The rates of participants determined to be MRD negative (MRD-) or positive for MRD (MRD+) will be reported as a percentage of participants.
Proportion of participants who produced adequate quantities of product for infusion | From initiation of BCMA CAR T-cell manufacturing to end of infusion, Up to 1 month
  To evaluate the feasibility of manufacturing anti-BCMA CAR T-cells locally and ability to produce adequate quantities of vector positive T-cells, the proportion of participants for whom BCMA CAR T-cell therapy is manufactured and meets pre-specified release criteria will be reported
Proportion of participants who complete Car-T infusion study treatment | From initiation of BCMA CAR T-cell manufacturing to end of infusion, Up to 1 month
  To evaluate the feasibility of manufacturing anti-BCMA CAR T-cells locally and ability to produce adequate quantities of vector positive T-cells, the proportion of participants successfully completed the BCMA CAR T-cell therapy is manufactured and meets pre-specified release criteria will be reported
Proportion of participants with treatment- emergent adverse events - Long Term | Up to 15 years
  The proportion of participants with treatment-emergent adverse events of CAR-T in RRMM, as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 5.0), revised CRS grading criteria (for CRS grading), and ASTCT ICANS Consensus Grading for Adults (for neurotoxicity grading) From initiation of BCMA CAR T-cell manufacturing to end of long-term follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Martin, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No